CLINICAL TRIAL: NCT04918251
Title: Investigation of EEG and TMS-based Biomarkers of Amyotrophic Lateral Sclerosis, Multiple Sclerosis and Frontotemporal Dementia
Brief Title: EEG and TMS-based Biomarkers of ALS, MS and FTD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Dublin, Trinity College (Other)
Collaborators: Motor Neurone Disease Association, UK (Unknown); Irish Research Council, IE (Unknown); Health Research Board, IE (Unknown); Research Motor Neurone, IE (Unknown); Thierry Latran Foundation, FR (Unknown); ALS Association, USA (Unknown)
Responsible Party: Principal Investigator, Orla Hardiman, Professor of Neurology, University of Dublin, Trinity College
Other Study IDs: CRFSJ00170; CRFSJ00171 (Other: St James' Hospital Clinical Research Facility, Dublin)
Record Dates: First submitted 2021-04-01; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Multiple Sclerosis
Keywords: EEG; TMS; Neurodegeneration; Network; Electrophysiology; Biomarkers; Cognitive; Behavioural; Motor
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Frontotemporal Dementia; Multiple Sclerosis; Nerve Degeneration | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Controls: Individuals from the Irish population with no psychiatric, psychological, neurological or muscular disease diagnosis
  Interventions: Procedure: 128 electrode electroencephalography (EEG); Procedure: Transcranial magnetic stimulation (TMS)
- Amyotrophic lateral sclerosis patients
  Interventions: Procedure: 128 electrode electroencephalography (EEG); Procedure: Transcranial magnetic stimulation (TMS)
- Multiple sclerosis patients
  Interventions: Procedure: 128 electrode electroencephalography (EEG); Procedure: Transcranial magnetic stimulation (TMS)
- Frontotemporal dementia patients
  Interventions: Procedure: 128 electrode electroencephalography (EEG); Procedure: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Procedure: 128 electrode electroencephalography (EEG) — 128 electrode EEG will be non-invasively recorded from electrodes placed in a montage over the scalp while the participant is resting or performing tasks designed to engage specific cortical motor networks of interest (cognitive, behavioural, motor and sensory)
Procedure: Transcranial magnetic stimulation (TMS) — Single and paired pulse TMS protocol will be delivered while surface bipolar EMG is recorded over hand muscles to interrogate corticospinal tract function and cortical motor network component functions

SUMMARY:
The purpose of this observational study is to improve understanding of the biology of why ALS, MS and FTD have different effects on different people and facilitate better measurement of the disease in future drug testing. To do this, brain and spinal cord neural network functionality will be measured over time, in addition to profiling of movement and non-movement symptoms, in large groups of patients, as well as in a population-based sample of the healthy population. Patterns of dysfunction which relate to patients' diagnosis and coinciding and future symptoms which align with categories of patients with similar prognoses will be investigated and their ability to predict incident patients' symptoms in future will be measured.

DETAILED DESCRIPTION:
The aim of this project is to characterize spatiotemporal patterns of central nervous system dysfunction that correlate with clinical features of ALS, MS and FTD, to provide non-invasive electrophysiological measurements that can be used in a clinical setting to inform stratification of patients in clinical trials, and to provide data driven diagnostic and prognostic biomarkers and objective clinical trial outcome measures. Such dysfunction will be investigated by recording single- and paired-pulse transcranial magnetic stimulation (TMS)-associated electromyography (EMG) during rest and by recording electroencephalography (EEG) during rest and during cognitive-motor tasks.

ELIGIBILITY:
Inclusion criteria:

* Age >18 years and able to give informed written or verbal (in the presence of two witnesses) consent.
* In the case of non-control subjects, a clinical diagnosis of:

  (i) Probable frontotemporal dementia (FTD) including behavioural variant FTD, semantic dementia or primary progressive aphasia) with supportive brain imaging or known FTD causing genetic mutation (ii) Multiple sclerosis (MS) according to the McDonald criteria (Polman et al., 2011) or (iii) Possible, probable or definite amyotrophic lateral sclerosis (ALS) according to the El Escorial Criteria Revised (Brooks et al. 2000)

Exclusion criteria:

* Any diagnosed neurological/muscular disease other than ALS, MS or FTD
* Use of neuro- or myo-modulatory medications except riluzole
* Inability to participate due to disease-related motor symptoms (e.g. inability to sit for the required time or click the mouse to respond)
* Upper body metallic implants
* History of seizure disorders in the participant or immediate family members
* Anxiety-induced fainting
* Regular migraine
* Evidence of significant respiratory insufficiency
* Sleep time >2 hours below normal and/or alcohol consumption the night before data collection (in which case, recording session will be rescheduled).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and patients diagnosed with ALS, FTD or MS
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Diagnosis-related difference in EEG or TMS measurements | Baseline recording
  Differences in single or paired pulse TMS measures or time and/or frequency domain EEG characteristics between those within each patient cohort and controls
Prognosis-related EEG or TMS measurements | Baseline recording
  Patient cohort single or paired pulse TMS measures or time and/or frequency domain EEG characteristics which show significant correlation to cognitive, behavioural, motor and/or sensory task performance, to disease duration or to survival time
Diagnosis-related changes in EEG or TMS measurements | Baseline to final visit assessed up to 2 years after baseline
  Differences in rate of change (slope) across time of single or paired pulse TMS measures or time and/or frequency domain EEG characteristics between those within each patient cohort relative to controls
Prognosis-related changes in EEG or TMS measurements | Baseline to final visit assessed up to 2 years after baseline
  Rates of change (slope) across time of patient cohort single or paired pulse TMS measures or time and/or frequency domain EEG characteristics which show significant correlation to cognitive, behavioural, motor and/or sensory task performance, to disease duration or to survival time

SECONDARY OUTCOMES:
Diagnosis-specific changes in EEG or TMS measurements | Baseline to final visit assessed up to 2 years after baseline
  Differences in rate of change (slope) across time of single or paired pulse TMS measures or time and/or frequency domain EEG characteristics between patient cohorts
Diagnosis-specific difference in EEG or TMS measurements | Baseline recording
  Differences in single or paired pulse TMS measures or time and/or frequency domain EEG characteristics between patient cohorts

CONTACTS AND LOCATIONS:
Overall Officials: Orla Hardiman, BSc MB BCh BAO MD FRCPI FAAN, Principal Investigator — Academic Unit of Neurology, Trinity College Dublin, The University of Dublin
Locations (1):
- Academic Unit of Neurology, Trinity College Dublin, The University of Dublin, Dublin, Leinster, Ireland

IPD SHARING:
Plan to Share IPD: Yes
Raw data from this study may be made available in anonymized form upon request from qualified investigators subject to the approval by the Data Protection Office (DPO) and Office of Corporate Partnership and Knowledge Exchanges (OCPKE) in Trinity College Dublin, the University of Dublin.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Due to ethical constraint and the time required for data quality checks, data will only be made available in fully anonymised format following publication of results.

REFERENCES:
- [Result] McMackin R, Dukic S, Broderick M, Iyer PM, Pinto-Grau M, Mohr K, Chipika R, Coffey A, Buxo T, Schuster C, Gavin B, Heverin M, Bede P, Pender N, Lalor EC, Muthuraman M, Hardiman O, Nasseroleslami B. Dysfunction of attention switching networks in amyotrophic lateral sclerosis. Neuroimage Clin. 2019;22:101707. doi: 10.1016/j.nicl.2019.101707. Epub 2019 Feb 2. PMID 30735860
- [Result] Dukic S, McMackin R, Buxo T, Fasano A, Chipika R, Pinto-Grau M, Costello E, Schuster C, Hammond M, Heverin M, Coffey A, Broderick M, Iyer PM, Mohr K, Gavin B, Pender N, Bede P, Muthuraman M, Lalor EC, Hardiman O, Nasseroleslami B. Patterned functional network disruption in amyotrophic lateral sclerosis. Hum Brain Mapp. 2019 Nov 1;40(16):4827-4842. doi: 10.1002/hbm.24740. Epub 2019 Jul 26. PMID 31348605
- [Result] McMackin R, Dukic S, Costello E, Pinto-Grau M, Fasano A, Buxo T, Heverin M, Reilly R, Muthuraman M, Pender N, Hardiman O, Nasseroleslami B. Localization of Brain Networks Engaged by the Sustained Attention to Response Task Provides Quantitative Markers of Executive Impairment in Amyotrophic Lateral Sclerosis. Cereb Cortex. 2020 Jul 30;30(9):4834-4846. doi: 10.1093/cercor/bhaa076. PMID 32318719
- [Result] McMackin R, Dukic S, Costello E, Pinto-Grau M, Keenan O, Fasano A, Buxo T, Heverin M, Reilly R, Pender N, Hardiman O, Nasseroleslami B. Sustained attention to response task-related beta oscillations relate to performance and provide a functional biomarker in ALS. J Neural Eng. 2021 Feb 25;18(2). doi: 10.1088/1741-2552/abd829. PMID 33395671
- [Result] Iyer PM, Mohr K, Broderick M, Gavin B, Burke T, Bede P, Pinto-Grau M, Pender NP, McLaughlin R, Vajda A, Heverin M, Lalor EC, Hardiman O, Nasseroleslami B. Mismatch Negativity as an Indicator of Cognitive Sub-Domain Dysfunction in Amyotrophic Lateral Sclerosis. Front Neurol. 2017 Aug 15;8:395. doi: 10.3389/fneur.2017.00395. eCollection 2017. PMID 28861032
- [Result] Nasseroleslami B, Dukic S, Broderick M, Mohr K, Schuster C, Gavin B, McLaughlin R, Heverin M, Vajda A, Iyer PM, Pender N, Bede P, Lalor EC, Hardiman O. Characteristic Increases in EEG Connectivity Correlate With Changes of Structural MRI in Amyotrophic Lateral Sclerosis. Cereb Cortex. 2019 Jan 1;29(1):27-41. doi: 10.1093/cercor/bhx301. PMID 29136131
- [Result] Iyer PM, Egan C, Pinto-Grau M, Burke T, Elamin M, Nasseroleslami B, Pender N, Lalor EC, Hardiman O. Functional Connectivity Changes in Resting-State EEG as Potential Biomarker for Amyotrophic Lateral Sclerosis. PLoS One. 2015 Jun 19;10(6):e0128682. doi: 10.1371/journal.pone.0128682. eCollection 2015. PMID 26091258